CLINICAL TRIAL: NCT02898818
Title: EMMI - Emättimen Mikrobiomi - Emättimen ja Suun Limakalvojen Vuorovaikutus
Brief Title: Vaginal and Oral Microbiome Crosstalk
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T146/2016
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Vaginal Discharge
MeSH Terms: conditions — Vaginal Discharge | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — swab sample from vaginal ja oral smear, including microbes and epithelial cells
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (5):
- symptomless: vaginal and oral swab sample, questionnaire
  Interventions: Other: vaginal and oral swab sample, questionnaire
- vaginal discharge: vaginal and oral swab sample, questionnaire
  Interventions: Other: vaginal and oral swab sample, questionnaire
- atypical papa smear: vaginal and oral swab sample, questionnaire, papa smear
  Interventions: Other: vaginal and oral swab sample, questionnaire; Other: papa smear
- no atypical papa smear: vaginal and oral swab sample, questionnaire, papa smear
  Interventions: Other: vaginal and oral swab sample, questionnaire; Other: papa smear
- lichen planus: vaginal and oral swab sample, questionnaire, papa smear
  Interventions: Other: vaginal and oral swab sample, questionnaire; Other: papa smear

INTERVENTIONS:
Other: vaginal and oral swab sample, questionnaire — vaginal and oral swab sample and questionnaire
Other: papa smear — Papnicolaou Papa Smear test
  Groups: atypical papa smear; lichen planus; no atypical papa smear

SUMMARY:
To study the vaginal and oral microbiome by swab samples. On selected cases, also papa smear will be studied.

DETAILED DESCRIPTION:
To study the vaginal and oral microbiome by swab samples and on selected groups, by papa smear test, to find out the constitution of normal and vaginal microbiome and the cross-talk between oral and vaginal mucosa. To find out about the impact of human papilloma virus on the microbiome and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* patients coming to Turku University Hospital Dermato-Venereology or Gynaecology Departments or to family planning clinics in The wellbeing services county of Southwest Finland for previously mentioned reasons

Exclusion Criteria:

* those not meeting the criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients coming to Turku University Hospital Dermato-Venereology Department for venereal disease tests with or without vaginal discharge. Patients coming to Turku University Hospital Gynaecology Department by remission because of atypical papa smear test result or (controls) for some other reason. Patients coming to family planning clinics in The wellbeing services county of Southwest Finland.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2017-04-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
microbiome, papa smear | 5 years
  Differences in microbiome and papa smear

CONTACTS AND LOCATIONS:
Overall Officials: Niina K Hieta, MD, PhD, Principal Investigator — specialist
Locations (1):
- Turku University Hospital, Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided